CLINICAL TRIAL: NCT05705141
Title: The Effect of Metabolic Syndrome on Antiviral Response in People With Chronic Hepatitis B: a Prospective, Multicenter, Real-world Study
Brief Title: The Effect of Metabolic Syndrome on Antiviral Response in People With Chronic Hepatitis B
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jie Li, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: CDL2302
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis b; metabolic syndrome; Antiviral treatment
MeSH Terms: conditions — Hepatitis B, Chronic; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined metabolic syndrome: HBeAg-positive CHB patients with metabolic syndrome
- Uncombined with metabolic syndrome: HBeAg-positive CHB patients without combined MS

SUMMARY:
Chronic hepatitis B (CHB) affects an estimated 292 million people, and causes approximately 800,000 people deaths per year from liver-related complications including cirrhosis and hepatocellular carcinoma, remaining a major global public health issue.Meanwhile, the rising incidence of metabolic syndrome (MetS) is another grim health burden. Combined MetS affects the metabolic function of hepatocytes, which are responsible for providing HBV replication. Antiviral therapy is an effective measure to reduce the risk of cirrhosis and liver cancer in patients with chronic CHB. Combined MetS may affect the antiviral efficacy in patients with CHB.This prospective observational study examines the differences in HBeAg serological conversion rates between HBeAg-positive CHB patients with and without MS who received first-line oral antivirals for 144 weeks.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) affects an estimated 292 million people, and causes approximately 800,000 people deaths per year from liver-related complications including cirrhosis and hepatocellular carcinoma, remaining a major global public health issue.Meanwhile, the rising incidence of metabolic syndrome (MetS) is another grim health burden. Combined MetS affects the metabolic function of hepatocytes, which are responsible for providing HBV replication. Antiviral therapy is an effective measure to reduce the risk of cirrhosis and liver cancer in patients with chronic CHB. Combined MetS may affect the antiviral efficacy in patients with CHB.This prospective observational study examines the differences in baseline clinical characteristics and the value of predicting HBeAg seroconversion rates at 144 weeks in HBeAg-positive CHB patients with and without MetS, and examines the differences in HBeAg seroconversion rates, degree of HBsAg decline, biochemical recurrence rates and HBV DNA negativity between HBeAg-positive CHB patients with and without MetS at 48 weeks, 96 weeks and 144 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender, age 18-65 years.
2. CHB diagnosis in accordance with the 2019 China Guidelines for the Prevention and Treatment of Chronic Hepatitis B; metabolic syndrome can be diagnosed with 3 or more of the following: 1) abdominal obesity: waist circumference ≥ 90 cm in men and ≥ 85 cm in women; 2) increased blood pressure: blood pressure ≥ 130/85 mmHg and/or diagnosed and treated hypertension; 3) dyslipidemia: fasting triglycerides ≥ 1.7 mmol/L, fasting HDL-C <1.04mmol/L, or diagnosed and medically treated dyslipidaemia; 4) Hyperglycaemia: fasting blood glucose ≥6.1mmol/L or 2 hours post sugar load blood glucose ≥7.8mmol/L, and/or diagnosed and treated diabetes mellitus.
3. HBeAg-positive, meeting the indications for antiviral treatment in our 2019 Guidelines for the Prevention and Treatment of Chronic Hepatitis B and ready to receive first-line antiviral medication.
4. voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients with co-infection with hepatitis A virus, hepatitis C virus, hepatitis E virus or hepatitis D virus
2. Patients with combined autoimmune hepatitis, primary biliary cholangitis or primary sclerosing cholangitis
3. Patients with co-morbid hereditary metabolic liver disease such as hepatomegaly, hepatic glycogen accumulation disorder
4. Patients with co-morbid primary liver cancer or other types of cancer; mental illness, severe cardiopulmonary impairment
5. Patients with alcohol abuse (≥210 g alcohol/week for men and ≥140 g alcohol/week for women)
6. Patients who have undergone liver transplantation or other organ transplantation.
7. Have received antiviral treatment within six months prior to enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-positive CHB patients with and without metabolic syndrome received first-line oral antiviral therapy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Difference of HBeAg seroconversion rate between HBeAg-positive CHB patients with and without metabolic syndrome after 144 weeks of first-line oral antiviral treatment | 144 weeks
  Difference of HBeAg seroconversion rate between HBeAg-positive CHB patients with and without metabolic syndrome after 144 weeks of first-line oral antiviral treatment

SECONDARY OUTCOMES:
Baseline clinical characteristics of HBeAg-positive CHB patients with and without metabolic syndrome, and the value of predicting HBeAg seroconversion rate at 144 weeks | 144 weeks
  Baseline clinical characteristics of HBeAg-positive CHB patients with and without metabolic syndrome, and the value of predicting HBeAg seroconversion rate at 144 weeks
Differences in rates of HBeAg seroconversion, HBsAg decline, biochemical relapse, and HBV DNA negativity between HBeAg positive CHB patients with and without metabolic syndrome treated for 48, 96, and 144 weeks | 48 weeks，96 weeks，144 weeks
  Differences in rates of HBeAg seroconversion, HBsAg decline, biochemical relapse, and HBV DNA negativity between HBeAg positive CHB patients with and without metabolic syndrome treated for 48, 96, and 144 weeks